CLINICAL TRIAL: NCT06747078
Title: The Effect of Core and Balance Exercises on Gait, Balance and Quality Of Life in Children With Cerebral Palsy: A Comparative Study
Brief Title: Comparison of Three Treatment in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hatice Özoymak Akçin, Principal Investigator MSc. Physiotherapist, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAU-FTR-HÖA-01
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy
Keywords: balance; Cerebral Palsy; Core Stabilization Exercise; Neurodevelopmental Therapy; Quality of life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Participants were divided into 3 groups. Group 1 (study group) received neurodevelopmental therapy (NDT) combined with core stabilization exercises (CSE). Group 2 (study group) received NDT combined with balance exercises (BE). The control group received only NDT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (study group): Neurodevelopmental therapy (NDT) combined with core stabilization exercises ( (Active Comparator): In addition to neurodevelopmental treatment, which is 30 minutes per day, 3 sessions per week and 24 sessions in total, core stabilization training was applied 3 sessions per week for 8 weeks and 24 sessions in total. The core stabilization training session lasted 30 minutes.
  Interventions: Other: Neurodevelopmental Therapy (NDT) + Core Stabilization Training
- Group 2 (study group) neurodevelopmental treatment combined with balance exercises (Active Comparator): In addition to the neurodevelopmental treatment of 30 minutes per day, 3 sessions per week, and a total of 24 sessions, balance training was applied 3 sessions per week for 8 weeks and a total of 24 sessions. The balance training session lasted 30 minutes.
  Interventions: Other: Neurodevelopmental therapy + Balance Exercises
- Group 3: Neurodevelopmental treatment control group (Active Comparator): Only neurodevelopmental treatment was applied for 60 minutes per day, 3 sessions per week, for 8 weeks, for a total of 24 sessions.
  Interventions: Other: Neurodevelopmental therapy

INTERVENTIONS:
Other: Neurodevelopmental Therapy (NDT) + Core Stabilization Training — In addition to the neurodevelopmental treatment of 30 minutes per day, 3 sessions per week, and a total of 24 sessions, core stabilization training was applied 3 sessions per week for 8 weeks and a total of 24 sessions. The core stabilization training session lasted 30 minutes.
  Other Names: NDT+CSE
  Arms: Group 1 (study group): Neurodevelopmental therapy (NDT) combined with core stabilization exercises (
Other: Neurodevelopmental therapy + Balance Exercises — In addition to NDT, which is 30 minutes per day, 3 sessions per week and 24 sessions in total, balance training was applied 3 sessions per week for 8 weeks and 24 sessions in total. The balance exercise session lasted 30 minutes.
  Other Names: NDT+BE
  Arms: Group 2 (study group) neurodevelopmental treatment combined with balance exercises
Other: Neurodevelopmental therapy — NDT was applied for 60 minutes per day, 3 sessions per week, for 8 weeks and a total of 24 sessions.
  Arms: Group 3: Neurodevelopmental treatment control group

SUMMARY:
In this study, considering the importance of walking and balance functions in improving the quality of life and achieving independence in children with cerebral palsy, it was aimed to examine whether core stabilization exercises specifically designed for children with cerebral palsy have an impact on improving balance and walking functions as well as quality of life. Additionally, the study sought to determine whether this approach has superiority over conventional balance exercises.

DETAILED DESCRIPTION:
Children with cerebral palsy included in the study were randomized into three groups using block randomization based on age, type of cerebral palsy and the Gross Motor Function Classification System (GMFCS). Children with cerebral palsy aged 7-18 years were included. Group 1 (study group, n=12) received neurodevelopmental therapy (NDT) combined with core stabilization exercises (CSE). Group 2 (study group, n=12) received NDT combined with balance exercises (BE). The control group (n=12) received only NDT. Treatments were conducted for 60 minutes per session, three times a week, over 8 weeks, for a total of 24 sessions, with an equal duration across groups. Participants' balance was evaluated using the Pediatric Balance Scale (PBS) and the SportKat 550® device. The Trunk Involvement Scale (TIS) was used to measure trunk impairment, the Six-Minute Walk Test (6MWT) to assess functional mobility and walking capacity and the Pediatric Outcome Data Collection Instrument (PODCI) to evaluate quality of life. All assessments were performed by the same physiotherapist before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Cases between the ages of 7-18
* Cases with GMFCS level I and II
* Cases diagnosed with hemiparetic and diparetic CP

Exclusion Criteria:

* Cases with levels III, IV and V according to GMFCS
* Having an intellectual disability that would prevent participation in assessment and exercise training
* Having had Botulinum Toxin (BOTOX) Type A application within the last 6 months
* Having undergone any surgical operation within the last 6 months
* Hearing and vision problems

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale (PBS) | eight weeks
  The Pediatric Balance Scale is used to assess functional balance skills in children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
SportKat550 Kinesthetic Ability Trainer (SportKAT 550) | eight weeks
  The SportKAT-550® device used to determine postural sway consists of sensors that detect sway and is also a balance platform. There is a digital screen in front of the platform to provide feedback to the person on it. The person on the platform is asked to hold the "X" mark on the digital screen in the center while the static balance test is performed. A score of 500 or lower than 500 in the static balance measurement indicates that the balance is good and the postural sway is low.For dynamic balance, a score between 750-950 is excellent, and a score between 1350-1550 indicates good balance.
Pediatric Outcome Data Collection Instrument (PODCI) | eight weeks
  It is a widely used scale to determine quality of life, functional health status and participation in children with cerebral palsy.The test is a Likert type scale and consists of 5 parts.PVTA, which has validity and reliability in Turkish, is scored between 0-100.

SECONDARY OUTCOMES:
Six Minute Walk Test (6MWT) | eight weeks
  The 6-minute walking test (6 MWT) is an easy test that is frequently used to determine functional mobility and walking distance in children with cerebral palsy. In our study, 6MWT was performed by measuring the distance the subject walked quickly but without running on a straight distance of 20 meters.
The Trunk Involvement Scale (TIS) | eight weeks
  The Trunk Involvement Scale was used to assess the trunk. It consists of three subsections: dynamic, static and coordination. Scoring can vary between 0-23.

OTHER OUTCOMES:
Gross Motor Function Classification System (GMFSS) | at the beginning of the study
  In our study, GMFCS was used to determine the gross motor functions of the subjects. This classification system is based on the movements initiated by the child by looking at sitting, moving and mobility. It consists of a five-level classification system.Level 1 and Level 2 children were included in the study

CONTACTS AND LOCATIONS:
Overall Officials: Nılufer CETISLI-KORKMAZ, PT.PhD.Prof, Study Director — Pamukkale University Faculty of Physiotherapy and Rehabilitation Block A
Locations (1):
- Pamukkale University Faculty of Physiotherapy and Rehabilitation Block A, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No